CLINICAL TRIAL: NCT03085368
Title: A Randomized Controlled Trial of HER-2 Positive Breast Cancer Patients Treated With Lapatinib and Paclitaxel vs Herceptin and Paclitaxel With Sequential and Synchronous Anthracycline
Brief Title: A Randomized Controlled Trial of HER-2 Positive Breast Cancer Patients Treated With Lapatinib vs Herceptin
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Taizhou EOC Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: lapatinib
Record Dates: First submitted 2017-03-19; First posted 2017-03-21 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: HER2-positive Breast Cancer
Keywords: breast cancer; her-2 positive; lapatinib; herceptin
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- EC→PL(Epirubicin+Cyclophosphamide--Docetaxel+lapatinib) (Experimental): Epirubicin 80 mg/ IV day M2 Cyclophosphamide 600 mg/m2 day IV 21 days for a total of 1 cycles, with a total of 4 cycles sequential Docetaxel 100mg/m2 IV day 1 21 days for a total of 1 cycles, with a total of 4 cycles Lapatinib 1000mg/d Po (fasting) every 30 days for a cycle Note: lapatinib in the first injection of docetaxel drug taking, once a day, oral dose of 1000mg, a total of over 1 years;
  Interventions: Drug: lapatinib/herceptin
- PEL(Paclitaxel+epirubicin+Lapatinib) (Experimental): 80mg/ M2 day 1 IV epirubicin Paclitaxel 150mg/m2 IV day 1 14 days for a total of 1 cycles (intensive chemotherapy), with a total of 6 cycles Also given Lapatinib 1000mg/d Po (fasting) every 30 days for a cycle Note: lapatinib in the first injection of paclitaxel drug taking, once a day, oral dose of 1000mg, a total of over 1 years;
  Interventions: Drug: lapatinib/herceptin
- EC→PH(Epirubicin+Cyclophosphamide--Docetaxel+herceptin) (Active Comparator): Table 80mg/ day 1 IV Cyclophosphamide 600 mg/m2 day IV 21 days for a total of 1 cycles, with a total of 4 cycles Docetaxel 100mg/m2 IV day 1 21 days for a total of 1 cycles, with a total of 4 cycles Trastuzumab 2mg/kg IV QW (first dose 4 mg/kg) Note: trastuzumab was administered at the beginning of the first injection of paclitaxel, with an injection dose of 2mg/kg, 1 times a week, for a total of up to 1 years; followed by trastuzumab 2mg/kg IV, once every 3 weeks for a total of one year
  Interventions: Drug: lapatinib/herceptin
- EPH(Paclitaxel+epirubicin+herceptin) (Active Comparator): 80mg/ M2 day 1 IV epirubicin Paclitaxel 150mg/m2 IV day 1 14 days for a total of 1 cycles, with a total of 6 cycles Also given Trastuzumab 2mg/kg IV QW (first dose 4 mg/kg) Note: trastuzumab was administered at the beginning of the first injection of paclitaxel, with an injection dose of 2mg/kg, 1 times a week, for a total of up to 1 years; followed by trastuzumab 2mg/kg IV, once every 3 weeks for a total of one year
  Interventions: Drug: lapatinib/herceptin

INTERVENTIONS:
Drug: lapatinib/herceptin — Lapatinib produced by glaxosmithkline. Oral small molecule epidermal growth factor tyrosine kinase inhibitor. Mainly used for combined with capecitabine in the treatment of ErbB-2 over expression, including received prior anthracycline, paclitaxel and trastuzumab (Herceptin) in the treatment of advanced or metastatic breast cancer. Our clinical trial want to see its benefit in early breast cancer

SUMMARY:
This is a randomized controlled trial of HER-2 positive breast cancer patients treated with lapatinib and paclitaxel vs herceptin and paclitaxel with sequential and synchronous anthracycline

DETAILED DESCRIPTION:
This is a randomized controlled trial of HER-2 positive breast cancer patients treated with lapatinib and paclitaxel vs herceptin and paclitaxel with sequential and synchronous anthracycline. Safety and efficacy are the primary endpoint. The positive expression of HER2 was confirmed by postoperative pathology in patients with breast adenocarcinoma (IDC). Patients who had not received any chemotherapy and targeted anti HER2 therapy.

In this study, the non inferiority design method, according to the wishes of patients and signed informed consent, randomly into the group, a total of 482 patients were enrolled in the trial group: the control group =1:1. The subjects were followed up for a total of 1 years, until the disease progressed, and the toxicity was not tolerated.

We want to study 84 months. The follow-up period was 5 years (the first adjuvant treatment time to the last follow-up) or the researchers decided to end the study.

ELIGIBILITY:
Inclusion Criteria:

1. the first diagnosis of invasive breast cancer, confirmed by histology or cytology, and surgical resection of the primary lesions before receiving any anti breast cancer treatment;
2. female patients, aged 18 years and less than 80 years of age;
3. surgical resection of the primary tumor pathological examination, showed HER2 positive (defined as immunohistochemistry [IHC] 3+ or fluorescence in situ hybridization (FISH) positive);
4. hormone receptor status is known, lymph node positive or sentinel lymph node negative but high risk factors
5. the eastern oncology cooperative group (ECOG) patients with physical status score was 0 -2;
6. baseline LVEF >50%
7. the relevant institutional review board (IRB) or independent ethics committee (IEC) written informed consent

Exclusion Criteria:

1. the subjects in pregnancy or lactation;
2. pregnant women may be within the first 7 days before pregnancy test positive (urine or serum).
3. received chemotherapy, endocrine or anti HER2 anti-tumor therapy;
4. congestive heart failure, unstable angina, heart failure or myocardial infarction and other diseases;
5. other invasive tumors (including the second primary breast cancer), may affect the outcome of the evaluation and program compliance; but the treatment of patients with disease free survival at least more than 5 years can be selected;
6. with chronic liver disease in patients with liver dysfunction and / or with clinical manifestations: the serum total bilirubin > 2.5 * ULN; or INR = 1.5 but no bilirubin. serum ALT or AST> * 3 * ULN; alkaline phosphatase >2.5 * ULN; ALT or AST can be gradually increased, but with gradually increasing fatigue, nausea and vomiting, fever, right upper quadrant pain or tenderness
7. hematopoietic dysfunction, defined as follows: neutrophil count (ANC) <1.5 * 109/L; platelet <100 * 109/L; hemoglobin <9 g/dL;
8. other serious diseases, including: congestive heart failure (heart function NYHA grade II, III, IV) or occurred within 6 months of congestive heart failure, unstable angina, arrhythmia, myocardial infarction patients can't control or other severe cardiovascular disease; breathing at rest or need oxygen therapy; serious infection; uncontrolled diabetes;
9. there is a serious psychological or mental abnormalities, estimated that the participants to participate in this study is not strong;
10. known to study drug allergy;
11. the past 30 days participated in the study of other drug clinical trials.

1, failed to complete the clinical trial of at least 1 cycles according to the program, can not carry out safety and efficacy evaluation 2, a serious violation of this research program, not in accordance with the prescribed dose, method and course of medication.

Patients will receive lapatinib treatment, until a predetermined end end point, or development of unacceptable toxicity, or withdrawal of consent, or illness or death, to appear before the subject.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
DFS | 3 years& 5 years
  Since the first randomized to disease recurrence or death occurred due to other reasons, the recurrence of the disease include local, regional, distant, ipsilateral or contralateral breast cancer (excluding breast lobular carcinoma in situ) and non malignant tumor secondary breast (except the skin basal cell carcinoma or squamous cell carcinoma, cervical cancer in situ cancer).

SECONDARY OUTCOMES:
OS | 5 years & 10 years
  0S is defined as the time from randomization to death due to any cause

OTHER OUTCOMES:
biomarker | 5 years
  A retrospective study was performed to examine the correlation between the prognosis of the two adjuvant and biomarkers, including but not limited to Ki67, PI3K, C-MYC, IGF1R, P95HER2, P53 and other biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Sun Qiang, M.D., Study Chair — PUMCH
Locations (1):
- PUMCH, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
After obtaining the primary endpoint, we will share our IPD

REFERENCES:
- [Result] Piccart-Gebhart M, Holmes E, Baselga J, de Azambuja E, Dueck AC, Viale G, Zujewski JA, Goldhirsch A, Armour A, Pritchard KI, McCullough AE, Dolci S, McFadden E, Holmes AP, Tonghua L, Eidtmann H, Dinh P, Di Cosimo S, Harbeck N, Tjulandin S, Im YH, Huang CS, Dieras V, Hillman DW, Wolff AC, Jackisch C, Lang I, Untch M, Smith I, Boyle F, Xu B, Gomez H, Suter T, Gelber RD, Perez EA. Adjuvant Lapatinib and Trastuzumab for Early Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer: Results From the Randomized Phase III Adjuvant Lapatinib and/or Trastuzumab Treatment Optimization Trial. J Clin Oncol. 2016 Apr 1;34(10):1034-42. doi: 10.1200/JCO.2015.62.1797. Epub 2015 Nov 23. PMID 26598744
- [Result] Goss PE, Smith IE, O'Shaughnessy J, Ejlertsen B, Kaufmann M, Boyle F, Buzdar AU, Fumoleau P, Gradishar W, Martin M, Moy B, Piccart-Gebhart M, Pritchard KI, Lindquist D, Chavarri-Guerra Y, Aktan G, Rappold E, Williams LS, Finkelstein DM; TEACH investigators. Adjuvant lapatinib for women with early-stage HER2-positive breast cancer: a randomised, controlled, phase 3 trial. Lancet Oncol. 2013 Jan;14(1):88-96. doi: 10.1016/S1470-2045(12)70508-9. Epub 2012 Dec 10. PMID 23234763